CLINICAL TRIAL: NCT06154382
Title: Eltroxin Administration to Patients With Extremely Low T4 Values in the Intensive Care Unit: Comparison Between Groups and Therapeutic Outcomes
Brief Title: Eltroxin Administration to Patients With Extremely Low T4 Values in the Intensive Care Unit
Status: Recruiting | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, sara dichtwald, Dr, Meir Medical Center
Other Study IDs: 0290-23-MMC
Record Dates: First submitted 2023-11-23; First posted 2023-12-04 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Thyroid; Functional Disturbance
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1: eltroxin administration: patients witn low T4 level who recieved eltroxin in ICU
  Interventions: Drug: Eltroxin administration
- group 2: no eltroxin administration: patients witn low T4 level who did not recieve eltroxin in ICU

INTERVENTIONS:
Drug: Eltroxin administration — eltroxin administration
  Groups: group 1: eltroxin administration

SUMMARY:
Nonthyroidal illness (formerly called sick euthyroid syndrome) is a common condition in patients hospitalized in the intensive care unit, and it is caused by changes in the levels of thyroid hormones in the blood . These changes are correlated to the severity of the critical illness, morbidity and mortality. This condition is characterized by low serum T3 levels, high rT3 levels, normal or low T4 levels, and normal or low TSH levels. Previous studies have shown a relationship between NTIS (nonthyroidal illness) and poor therapeutic outcomes in patients admitted with sepsis, multi trauma, ARDS, acute respiratory failure, septic shock and mechanically ventilated patients in intensive care .

In general, the recommendation is not to routinely take blood tests to evaluate thyroid function in critical patients in the intensive care unit, unless they were previously known to have a thyroid disease or there is a clinical suspicion that such a disorder developed during hospitalization in the intensive care unit. Also, studies so far have not shown an advantage for eltroxin administration to intensive care patients with low T3 and/or T4 levels when the laboratory tests indicate NTIS. However, there is a specific group of patients, with NTIS and extremely low T4 levels (less than 50% of the lower limit of the normal range) who have a particularly high mortality rate in intensive care (over 85%) and in whom it has not been investigated whether the administration of eltroxin will improve the therapeutic outcomes ( , i.e. was such a low T4 level in them considered a marker for the severity of their general critical illness, or is it another disorder in itself, the treatment of which would benefit the patient) . We would like to examine whether the administration of eltroxin in this specific group of patients, which has not been studied so far, will be beneficial in improving the therapeutic outcomes

ELIGIBILITY:
Inclusion Criteria: All patients aged 18--99 who were admitted to the general intensive care unit from January 2016 to November 22, 2023 for any reason, and who during their hospitalization in the intensive care unit had lower than normal T4 levels measured. It is about 350 patients. Of these, we will specifically examine the group of patients for whom an extremely low level of T4 was measured (less than 50% of the lower limit of the norm).

-

Exclusion Criteria: Patients who were known to have a chronic thyroid dysfunction prior to their hospitalization in the unit, patients who were regularly treated with eltroxin prior to their hospitalization

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged 18--99 who were admitted to the general intensive care unit from January 2016 to November 22, 2023 for any reason, and who during their hospitalization in the intensive care unit had lower than normal T4 levels measured. It is about 350 patients. Of these, we will specifically examine the group of patients for whom an extremely low level of T4 was measured (less than 50% of the lower limit of the norm).
  -
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | 28-day mortality
  To examine whether there are differences in mortality within 28 days in intensive care patients with NTIS and extremely low levels (less than 50% of the lower limit of normal) of T4 between a group of patients who received eltroxin and another who did not.

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No